CLINICAL TRIAL: NCT04261114
Title: Exploring the Relationship Between Physical Pain and Emotional Distress in Adolescents with Chronic Pain - a Three-step Observational Follow-up Study
Brief Title: Exploring the Link Between Pain and Distress in Adolescent Patients with Chronic Pain
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Oskar-Helene-Heim Foundation (Other)
Responsible Party: Principal Investigator, VerenaHinze, Principal Investigator, University of Oxford
Other Study IDs: PID14553-SP001-AC001
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Adolescents; Emotional distress; Burdensomeness; Self-harm; Hopelessness
MeSH Terms: conditions — Chronic Pain; Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary aim is to explore what it is about the experience of chronic pain that may cause emotional distress in some young people but not in others, and how particular individual characteristics, as well as family factors may contribute to young persons' pain experiences and their emotional responses to pain.

DETAILED DESCRIPTION:
This is a three-part observational follow-up study:

Part one will explore (a) whether the current sample reports emotional distress, including feelings of burdensomeness, hopelessness and thoughts and acts of self-harm, and if young people perceive there to be a link between pain and any such feelings of distress, and (b) which aspects of the pain experience, if any, are associated with such distress, using qualitative and quantitative data.

Part two will explore potential individual-level and family-level risk and resilience factors underpinning the hypothesised relationship between aspects of the pain experience and burdensomeness, hopelessness and thoughts and acts of self-harm, using adolescent and parental baseline data.

In part three, adolescent participants will be invited to complete daily diaries on their pain experience, three times per day over 7 days, in order to investigate which aspects of the pain experience are associated with burdensomeness and hopelessness at follow-up.

This study has the potential to improve the care of young people with chronic pain, and in particular the emotional support that young people receive.

ELIGIBILITY:
Inclusion Criteria:

Part 1: Adolescents

* Participant is willing and able to give assent (aged 12-15) or informed consent (aged =>16) for participation in the study
* Adolescents aged 12 to 19 years
* Self-reported experience of chronic pain (i.e., recurrent and/or persistent pain at least once per week for at least 3 months).
* Able to read and converse fluently in English
* Parent/carer willing to give informed consent for participants aged 12-15

Part 2: Adults

* Participant is willing and able to give informed consent for participation in the study.
* Participant is the parent/carer for a child aged 12 to 19 years, with chronic pain (i.e., recurrent or persistent pain at least once per week for the past 3 months), and this child is participating in this study.
* Able to read and converse fluently in English

Additional criteria for Part 3: Follow-up part

· In possession of a smartphone to complete the momentary assessments.

Exclusion Criteria:

Part 1: Adolescents

* If some type of serious pathology (e.g., infection, fracture, disease process (e.g., cancer)) or surgical procedure is the cause of the resulting pain complaint.
* If the patient is too psychologically unstable (e.g., experience of hallucinations or delusions, or with known acute suicide risk) to safely participate in this research, based on clinical judgment.

Part 2: Adults

-If the clinical care team thinks the parent/ caregiver is unsuitable for this study.

Additional criteria for Part 3: Follow-up part

-Inability to provide data via the use of a smartphone

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 77 Adolescents with chronic pain and their parents/ caregivers
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Perceived burdensomeness | at baseline
  Interpersonal Needs Questionnaire (INQ), completed by the adolescents. Scores range from 1="not at all true for me" to 7="very true for me", with higher scores indicating more perceived burdensomeness.

SECONDARY OUTCOMES:
Perceived burdensomeness | at 7-day follow-up
  Interpersonal Needs Questionnaire (INQ), completed by the adolescents. Scores range from 1="not at all true for me" to 7="very true for me", with higher scores indicating more perceived burdensomeness.
Hopelessness | at baseline
  Hopelessness Scale for Children (HSC), completed by the adolescents. Participants score each item as 1=True and 0=False. The higher the score, the greater the hopelessness for the future.
Hopelessness | at 7-day follow-up
  Hopelessness Scale for Children (HSC), completed by the adolescents. Participants score each item as 1=True and 0=False. The higher the score, the greater the hopelessness for the future.
Thoughts and acts of self-harm | at baseline
  4 single items on the presence/ absence of self-harm thoughts and acts, completed by the adolescents.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Centre for Children and Young People in Pain, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The syntax code and a fully de-identified version of the final dataset may be shared with third parties to support future related research where it is in the public interest.